CLINICAL TRIAL: NCT03401931
Title: Artificial Intelligence Use for the Detection of Atrial Fibrillation Drivers
Acronym: AI Fib
Status: Withdrawn | Type: Observational
Why Stopped: another design of protocole is submitted for approuval before the start date
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Principal Investigator, SEITZ JULIEN, Cardiologist, Electrophysiology specialist, Hospital St. Joseph, Marseille, France
Other Study IDs: HSJ_AIFIB_2017
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Fibrillation, Atrial; To Evaluate the Intraoperative Efficiency of the AIFIB Software in the Detection of Atrial Fibrillation Driver During an Ablation Procedure
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
pilot clinical study, multicenter, prospective, open, nonrandomized

DETAILED DESCRIPTION:
The hypothesis is that ablation targeting PVI alone for the treatment of persistent AF is less efficient that ablation targeting electrophysiologic areas with spatio-temporal-dispersion with or without PVI

ELIGIBILITY:
Inclusion Criteria: major patient with an indication of AF or AT ablation -

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: major patient with an indication of AF or AT ablation
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2018-01-09 (Actual); Study Completion 2018-01-09 (Actual)

PRIMARY OUTCOMES:
AF termination | during the ablation procedure
  conversion to sinus rhythm or stable atrial tachycardia

SECONDARY OUTCOMES:
AT termination | during the ablation procedure
  conversion to sinus rhythm

CONTACTS AND LOCATIONS:
Overall Officials: Julien SEITZ, MD, Principal Investigator — Hopital saint Joseph
Locations (3):
- France (2):
  - Hopital d'Aix en Provence, Aix-en-Provence
  - CHU Nice, Nice
- Isala Hospital, Zwolle, Netherland, Netherlands